CLINICAL TRIAL: NCT06041048
Title: Investigation of Locus Coeruleus Function in Sustained Attention
Acronym: LC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1939774
Record Dates: First submitted 2023-07-17; First posted 2023-09-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Attention - no Condition is Being Assessed - Healthy Adults
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modafinil (Active Comparator): Single oral dose (200 mg) of medication versus placebo given to healthy control subjects
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Single dose (200 mg) of medication versus placebo given to healthy control subjects
  Other Names: Provigil

SUMMARY:
The norepinephrine-producing locus coeruleus (LC) is thought to be central to a wide array of cognitive functions, like attention and goal pursuit, and has been implicated in dysfunctions including attention deficit hyperactivity disorder and schizophrenia. The goal of this proposal is to develop methods that permit measurement of activity in the human LC. Because the LC is small and located in the pons, the Investigators will use high resolution magnetic resonance imaging techniques tailored to the brainstem environment, including neuromelanin-sensitive images shown to delineate the LC, combined with pharmacological manipulation to confirm the location of functional activity.

DETAILED DESCRIPTION:
Attention failures negatively impact goal pursuit and have significant consequences on performance in many environments. Attentional control of perceptual, motor and cognitive functions are believed to be partly determined by functioning of the locus coeruleus-norepinephrine (LC-NE) system. The LC, a small brainstem nucleus that is the primary source for NE in the forebrain, has motivated hypotheses about human cognition, including mental health disorders with known alterations in attention and cognition (e.g., attentiondeficit/ hyperactivity disorder (ADHD), schizophrenia) even though methods for measuring human LC activity have significant limitations. Existing methods to study LC function in humans rely on pupillometry and fMRI.

Because pupil diameter correlates with LC activity, it has been used as a proxy for LC activity. However, the anatomical pathway linking the LC to pupil dilation has not been established and pupil diameter also correlates with activity in other brain areas. Thus, inferring LC activity from pupillometry alone is problematic. fMRI has also been used to measure activity from the LC, but the imaging methods used to date have relied on resolutions that are coarse relative to the size and shape of LC. Prior fMRI results have therefore not been adequate for event-related analyses. The goal of the proposed work is to develop and validate methods for using fMRI to measure LC activity, specifically event-related responses that will allow for testing of influential hypotheses of LC function in humans. This goal is appropriate for the R21 mechanism, which is meant to "encourage exploratory/developmental research by providing support for the early and conceptual stages of project development" and to test innovative, high-risk, high reward research. This project has two specific aims, which are both tested with sustained attention tasks. The first aim uses high-resolution fMRI to maximize the number of measurements within LC combined with neuromelanin-sensitive imaging to localize BOLD responses to LC. The Investigators will measure (a) pre-trial activity (i.e., during inter-trial intervals; this period is thought to reflect tonic LC activity) and (b) trial response (i.e., phasic LC activity) by estimating the beta weights for each trial. The second aim uses modafinil administration to modulate LC activity and confirm the location of BOLD responses measured during the sustained attention tasks to the LC. The Investigators will administer modafinil and placebo to participants in a double-blind, placebo-controlled crossover study. Pupillometry data will also be collected for both the modafinil and placebo conditions, and the Investigators will use the pupillometry data to test for a correlation with LC BOLD response amplitude. This combination of techniques will demonstrate whether fMRI can be used to measure LC activity in a targeted fashion. Developing these tools meets Goal 1 (Strategy 1.3D) of the 2020 Strategic Plan of the NIMH by permitting direct measurement of a brain structure central in attentional control.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 - 60 years of age,
* Typically developing, healthy adult

Exclusion Criteria:

* History of schizophrenia, other forms of psychosis,
* Specific or focal neurological disorder or severe alcohol or drug use disorder within the past 5 years
* History of left ventricular hypertrophy or in patients with mitral valve prolapse who have experienced the mitral valve prolapse syndrome when previously receiving CNS stimulants, or who have had recent history of myocardial infarction or unstable angina.
* Volunteers with known hypersensitivity to modafinil or armodafinil or its inactive ingredients
* Known allergy/sensitivity or any hypersensitivity to components of modafinil or its formulation
* Inability to swallow tablets or tolerate oral medication;
* Pregnant or nursing (participants will be required to have a negative pregnancy test)
* Contraindication for MRI scanning (metal implants, pacemakers, metal foreign bodies, or pregnancy)
* Use of psychotropic medication within the past week
* Claustrophobic and not comfortable being in a small space may also not want to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Brain activity - BOLD response | 1 hour

SECONDARY OUTCOMES:
Attention on Oddball and POP task | 1 hour
  Response time and accuracy on Oddball and POP task

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded to the NIH NDA, following their procedures.
Supporting Information: Study Protocol
Time Frame: Within two years after data are analyzed by the investigative team. How long it will be available is determined by the NIH.